CLINICAL TRIAL: NCT00829205
Title: A Phase I/II Study of Methylselenocysteine (MSC) in Combination With Immunochemotherapy (R-ICE) in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Se-Methyl-Seleno-L-Cysteine, Rituximab, Ifosfamide, Carboplatin, and Etoposide in Treating Patients With Diffuse Large B-Cell Lymphoma That Has Relapsed or Not Responded to Treatment
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000632722; CRUK-UCL-SelRICE; EUDRACT-2008-002678-36; EU-20902
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-07

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Filgrastim; Rituximab; selenomethylselenocysteine; Carboplatin; Etoposide; Ifosfamide

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Dietary Supplement: Se-methyl-seleno-L-cysteine
Drug: carboplatin
Drug: etoposide
Drug: ifosfamide
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer cell-killing substances to them. Drugs used in chemotherapy, such as ifosfamide, carboplatin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Se-methyl-seleno-l-cysteine may help reduce the side effects of chemotherapy.

PURPOSE: This phase I/II trial is studying the side effects and best dose of Se-methyl-seleno-l-cysteine when given together with rituximab, ifosfamide, carboplatin, and etoposide and to see how well it works in treating patients with diffuse large B-cell lymphoma that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess dose-limiting toxicity and maximum-tolerated dose (MTD) of Se-methyl-seleno-L-cysteine (MSC) (to achieve a trough serum selenium [Se] concentration of > 20 μmol/L) prior to and in combination with rituximab, ifosfamide, carboplatin, and etoposide (R-ICE) in patients with relapsed or refractory diffuse large B-cell lymphoma. (Phase I)
* To determine the overall response rate to R-ICE given in addition to MSC at the MTD in these patients. (Phase II)

Secondary

* To determine the toxicity of R-ICE when used in combination with MSC in these patients.
* To determine the effect of MSC dosing on serum and intracellular Se and Se species in these patients.
* To determine the pharmacokinetics of MSC after single and multiple daily dosing in these patients.
* To investigate the effect of MSC dosing on Se-dependent processes (e.g., NFκB activity and AKT).

OUTLINE: This is a multicenter, phase I, dose-escalation study of Se-methyl-seleno-L-cysteine (MSC) followed by a phase II study.

Patients receive rituximab IV on day 1, carboplatin IV on day 2, ifosfamide IV and etoposide IV on days 2-4 (R-ICE), and filgrastim (G-CSF) subcutaneously on days 6-13. Patients also receive oral MSC twice daily on days -7 to 0 and once daily in courses 1-2. Treatment with R-ICE and G-CSF repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically and analyzed for pharmacokinetics and protein markers.

After completion of study treatment, patients are followed monthly for 3 months.

This study is peer reviewed and funded or endorsed by cancer research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed, CD20+, diffuse large B-cell lymphoma (DLBCL) according to WHO lymphoma classification

  * Histological transformation of a previously known indolent lymphoma allowed
  * Biopsy-proven DLBCL arising from an indolent lymphoma not diagnosed previously allowed
* Disease in first relapse after complete remission, partial response (PR), or less than a PR after first-line of treatment
* No primary CNS lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Serum creatinine < 150 μmol/L
* Serum bilirubin < 35 μmol/L
* Transaminases < 2.5 times upper limit of normal (unless attributed to lymphoma)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindication to any of the drugs contained in the immunochemotherapy regimen
* No other malignancy within the past 2 years, except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* No other serious active disease that, in the opinion of the investigator, would preclude the patient from having conventional chemotherapy
* No HIV positivity
* No medical or psychiatric conditions that compromise the patient's ability to give informed consent

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose of Se-methyl-seleno-L-cysteine (MSC) (Phase I)
Overall response rate (Phase II)

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v 3.0
Serum and intracellular Se and Se species
Pharmacokinetics of MSC
Protein markers of selenium activity

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Montoto, MD, Principal Investigator — Barts and the London NHS Trust
Locations (5):
- United Kingdom (5):
  - Barts and the London NHS Trust, London, England
  - Saint Bartholomew's Hospital, London, England
  - Christie Hospital, Manchester, England
  - Derriford Hospital, Plymouth, England
  - Southampton General Hospital, Southampton, England